CLINICAL TRIAL: NCT05761678
Title: Quality of Life of Transgender People - Implementation and Monitoring of an Online Cohort
Brief Title: Quality of Life of Transgender People - Implementation and Monitoring of an Online Cohort (e-QoL-Trans)
Acronym: e-QoL-Trans
Status: Recruiting | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A03156-35
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Transgenderism; Gender Identity
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender people: Whether they have transitioned or not, with or without reassignment surgery.
  Interventions: Other: Questionnaire quality of life

INTERVENTIONS:
Other: Questionnaire quality of life — Quantitative - Validated online self-questionnaires scientifically to assess quality of life and support perceived social. Items created for the study concerning socio-demographic characteristics and satisfaction of health services concerning the accompaniment of the transidentity.
  Qualitative - Semi-structured interviews based on a guide maintenance.

SUMMARY:
Transgender people have an identity or an expression gender that differs from the sex assigned to them at the birth. Transgender people and their needs remain misunderstood, and more generally by society. THE transgender populations express poor quality of life compared to the general population. However, very few of studies are interested in these people, in their diversity of paths, trajectories and characteristics of life. More of research is needed to study the quality of life, understand the experiences, in their diversity and in the health, social and life trajectories. Researches must be carried out, in particular on how to interrogate by the seeks out transgender people, in order to prevent stigmatization within population studies.

The main objective of this study is to assess the quality of life of people transgender people during their life trajectory and their transition path, based on validated questionnaires scientifically in French, for major themes of the population concerned (quality of life, social support perceived).

ELIGIBILITY:
Inclusion Criteria:

* Transgender people (having a gender identity or expression that differs from the sex assigned to them at birth);
* People with any of the following characteristics regarding their trans identity:

  * Consultant in one of the transgender reference centers and services for questions/information on the transition;
  * Integrated or having completed a course of care with or without gender reassignment surgery;
  * Not integrated into a health or care pathway.
* French-speaking people;
* Adults;
* People able to use the tools digital;
* People with Internet or 4G access (total or limited)

Exclusion Criteria:

* People who do not identify as transgender;
* Non-French speaking people;
* Minors
* People who do not know how to handle the tools digital data collection;
* People without Internet access.
* Non-French speaking people, unable to speak understand the research questions
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by court order or administrative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender people (having a gender identity or expression that differs from the sex assigned to them at birth)
Study Population: Transgender people, whether they have transitioned or not, with or without reassignment surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Quality of life estimated with a validated questionnaire administered over the Internet repeatedly every three months. | 3 months
  Quality of life estimated with a validated questionnaire administered over the Internet repeatedly every three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé Jean Mermoz, Lyon, France